CLINICAL TRIAL: NCT03169517
Title: Blood Flow Index as an Indicator of Successful Peripheral Nerve Block : A Prospective Observational Study Using Laser Speckle Contrast Imaging.
Brief Title: Blood Flow Index as an Indicator of Successful Peripheral Nerve Block
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Vice Director, Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: TJMZK20170325
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Laser
Keywords: Peripheral nerve block; laser speckle contrast imaging; blood flow index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral nerve block group: patients scheduled for elective upper or lower limb surgery with peripheral nerve block will receive LSCI measurements and pinprick sensory tests at 5 min before the block and at 5-min intervals till 30 min after the block.

SUMMARY:
Laser speckle contrast imaging (LSCI) allows real-time, non-invasive, quantitative measurements of regional blood flow. The aim of this prospective observational study was to evaluate the blood flow changes by LSCI after peripheral nerve block and determine whether this novel optical technique can be used as a reliable indicator of successful blocks.

DETAILED DESCRIPTION:
Methods: One hundred adult patients scheduled for elective upper or lower limb surgery with peripheral nerve block will receive LSCI measurements and pinprick sensory tests before the block and at 5-min intervals till 30 min after the block. The sensitivity, specificity of LSCI as a diagnostic method will be determined by receiver operator characteristic analysis.

Clinical Implications: LSCI with quantitative data could be used as an indicator of successful blocks.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* American Society of Anesthesiologists physical statusⅠ-Ⅱ
* Undergo elective upper or lower limb surgery with peripheral nerve block

Exclusion Criteria:

* refusal to participate in the study
* peripheral vascular disease
* digit injury or deficiency
* colored or infected fingernails/toenails
* BMI>35
* those who had taken vasodilatory drugs before surgery
* preoperative analgesic medications
* Any contraindications to peripheral nerve block such as coagulation abnormalities, allergy to local anaesthetics, peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: One hundred adult patients scheduled for elective upper or lower limb surgery with peripheral nerve block
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
diagnostic power of LSCI and pinprick sensory tests for predicting successful and failed blocks | at 5-min intervals till 30 min after regional block
  sensitivity and specificity

SECONDARY OUTCOMES:
blood flow index | 5 min before regional block and at 5-min intervals till 30 min after regional block
  perfusion unit(PU)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
For patient's privacy

REFERENCES:
- [Derived] Wu X, Li J, Joypaul K, Bao WW, Wang D, Huang YJ, Li PC, Mei W. Blood flow index as an indicator of successful sciatic nerve block: a prospective observational study using laser speckle contrast imaging. Br J Anaesth. 2018 Oct;121(4):859-866. doi: 10.1016/j.bja.2018.05.065. Epub 2018 Jul 4. PMID 30236247